CLINICAL TRIAL: NCT03876808
Title: A Prospective Randomized Clinical Trial Evaluating the Effect of Convective Pre-warming on Intra-operative Thermoregulatory Capabilities in Patients Enrolled in the TIGER Anesthesia Perioperative Protocol
Brief Title: The Effect of Convective Pre-warming on Intra-operative Thermoregulatory Capabilities
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor participant recruitment
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Boris Mraovic, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008755
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Temperature Change, Body
Keywords: temperature; prewarming; convective warming; thermoregulation; gastrointestinal surgery; genitourinary surgery
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Masking Description: At time of consent the randomization is masked for the participant, care provider, and investigator. Once randomization has occurred there is no masking as you clearly know what group has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Convective pre-warming (Experimental): Undergo convective warming during the preoperative preparations, completed for a minimum of 60 minutes prior to entering the operating room
  Interventions: Device: Bair Hugger™ Temperature Management Unit Model 750; Device: 3M™ Bair Paws™ Flex Gown
- Standard of care (No Intervention): Undergo standard of care, which includes providing each patient with blankets and sheets, as well as more blankets on patient request.

INTERVENTIONS:
Device: Bair Hugger™ Temperature Management Unit Model 750 — Forced-air temperature management unit used for preoperative and intraoperative participant warming
  Arms: Convective pre-warming
Device: 3M™ Bair Paws™ Flex Gown — Bair Paws™ patient warming gown used for preoperative and intraoperative participant warming
  Arms: Convective pre-warming

SUMMARY:
This prospective randomized clinical trial will assess the effect of pre-operative convective warming on intra-operative thermoregulation in patients undergoing gastrointestinal or genitourinary surgical procedures with the Tiger anesthesia perioperative protocol.

DETAILED DESCRIPTION:
By the year 2030 the geriatric presence in the United States, defined as any adult >65 years of age, is estimated to reach around 20% of the entire population. Thus, understanding medical concepts as they relate to the elderly is becoming increasingly important. One such concept is that of hypothermia - a core body temperature < 36°C - for which age >65 has been found to be an independent risk factor. This complication is especially prevalent intra-operatively due to use of general anesthetics, cool ambient operating room (OR) temperatures, and impaired thermal regulation in the elderly.

The human body employs numerous mechanisms to maintain thermal homeostasis including: behavioral means of thermoregulation, sweating, pre-capillary vasodilation, non-shivering and shivering means of heat production, and arteriovenous shunt vasoconstriction. The first, and arguably most important, regulatory response to occur is that of vasoconstriction, which normally results in redistribution of blood from the relatively cool periphery to the warmer core compartment in order to confine metabolic heat to the central tissues. Patients undergoing general anesthesia experience reduced vasoconstriction due to decreased cold response thresholds while patients undergoing epidural anesthesia experience sympathetic blocks resulting in blunted vasoconstrictive responses. All patients experience the afore mentioned side effects of anesthetics, however it has been proven that the elderly are more susceptible to hypothermia due to lower vasoconstriction thresholds - determined by a temperature gradient of 4°C between the periphery and core.

First explored by Kurz et al. in 1993, it was found that use of nitrous oxide and isoflurane anesthesia lead to an approximately 1.2°C lower vasoconstriction threshold of 33.9±0.6 in the elderly versus 35.1±0.3 in the young (p < .01). This subject was again looked at in a 1997 study wherein the vasoconstriction threshold during nitrous oxide and sevoflurane was observed to be decreased by approximately 0.8°C in the elderly at 35.0±0.8 versus 35.8±0.3 in the young (p < .01). This is relevant because intraoperative hypothermia has long been known to lead to adverse outcomes such as increased incidence of myocardial ischemia, arrhythmias, coagulopathic states, and wound infections. In a 2014 retrospective cohort study by Billeter et al. patient's experiencing core temperatures <35°C had a four times increase in mortality with complication rates increasing two fold and incidence of stroke increasing six fold. To counter this thermoregulatory failure in patients, numerous methods of warming have been practiced over time to augment the normal body response.

One method used to decrease intraoperative hypothermia is warming patients before surgery via skin surface warmers. Numerous studies have found that even brief periods of pre-warming can improve intraoperative temperatures significantly for as long as 75-90 minutes after induction. In procedures lasting less than 90 minutes, Horn et al. found that as little as 10 minutes of pre-warming decreased incidence of intraoperative hypothermia from 69% to just 13% while Torossian et al. decreased the incidence from 60% to 38% in his study using a self-warming blanket for 30 minutes pre-operatively. Studies have also shown that longer pre-warming, of 45-60 minutes, can prevent hypothermia for up to 2 hours after induction.

While significant research has been performed on the effects of warming patients before they undergo surgical procedures, scant evidence demonstrates the effect of pre-warming in the elderly. In one article specifically looking at pre-warming in the elderly (mean age ~72-73) it was found that, after pre-warming for 20 minutes, there was no significant change in incidence of hypothermia but there was a significant difference in severity of hypothermia when it did occur. This study focused only on men undergoing transurethral resection of the prostate however, and suffers from lack of generalizability. With the proportion of the geriatric population continuing to expand, and the potential adverse effects resulting from their increased susceptibility to intraoperative hypothermia, it is of the utmost importance to look into methods to counter this dilemma and expand the database on the topic.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-IV
* Other inclusion criteria as delineated in the TIGER anesthesia perioperative protocol

Exclusion Criteria:

* Inability to obtain written informed consent
* Inability to obtain core body temperature recordings
* Family history of malignant hyperthermia
* Preoperative temperature > 38° C
* Other exclusion criteria as delineated in the TIGER anesthesia perioperative protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Mraovic, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. The state of aging and health in America 2013. Atlanta, GA: Centers for Disease Control and Prevention, US Department of Health and Human Services, 2013.
- [Background] Billeter AT, Hohmann SF, Druen D, Cannon R, Polk HC Jr. Unintentional perioperative hypothermia is associated with severe complications and high mortality in elective operations. Surgery. 2014 Nov;156(5):1245-52. doi: 10.1016/j.surg.2014.04.024. Epub 2014 Jun 16. PMID 24947647
- [Background] Frank SM, Beattie C, Christopherson R, Norris EJ, Rock P, Parker S, Kimball AW Jr. Epidural versus general anesthesia, ambient operating room temperature, and patient age as predictors of inadvertent hypothermia. Anesthesiology. 1992 Aug;77(2):252-7. doi: 10.1097/00000542-199208000-00005. PMID 1642343
- [Background] Sessler, Daniel I. Chapter 8: preoperative thermoregulation. Geriatric Anesthesia, 2nd ed., Springer, New York, NY: 107-118, 2008.
- [Background] Glosten B, Hynson J, Sessler DI, McGuire J. Preanesthetic skin-surface warming reduces redistribution hypothermia caused by epidural block. Anesth Analg. 1993 Sep;77(3):488-93. doi: 10.1213/00000539-199309000-00012. PMID 8368549
- [Background] Kurz A, Plattner O, Sessler DI, Huemer G, Redl G, Lackner F. The threshold for thermoregulatory vasoconstriction during nitrous oxide/isoflurane anesthesia is lower in elderly than in young patients. Anesthesiology. 1993 Sep;79(3):465-9. doi: 10.1097/00000542-199309000-00008. PMID 8363070
- [Background] Ozaki M, Sessler DI, Matsukawa T, Ozaki K, Atarashi K, Negishi C, Suzuki H. The threshold for thermoregulatory vasoconstriction during nitrous oxide/sevoflurane anesthesia is reduced in the elderly. Anesth Analg. 1997 May;84(5):1029-33. doi: 10.1097/00000539-199705000-00014. PMID 9141926
- [Background] Kim JY, Shinn H, Oh YJ, Hong YW, Kwak HJ, Kwak YL. The effect of skin surface warming during anesthesia preparation on preventing redistribution hypothermia in the early operative period of off-pump coronary artery bypass surgery. Eur J Cardiothorac Surg. 2006 Mar;29(3):343-7. doi: 10.1016/j.ejcts.2005.12.020. Epub 2006 Jan 24. PMID 16434206
- [Background] Perl T, Peichl LH, Reyntjens K, Deblaere I, Zaballos JM, Brauer A. Efficacy of a novel prewarming system in the prevention of perioperative hypothermia. A prospective, randomized, multicenter study. Minerva Anestesiol. 2014 Apr;80(4):436-43. Epub 2013 Oct 3. PMID 24193180
- [Background] Horn EP, Bein B, Bohm R, Steinfath M, Sahili N, Hocker J. The effect of short time periods of pre-operative warming in the prevention of peri-operative hypothermia. Anaesthesia. 2012 Jun;67(6):612-7. doi: 10.1111/j.1365-2044.2012.07073.x. Epub 2012 Feb 29. PMID 22376088
- [Background] Torossian A, Van Gerven E, Geertsen K, Horn B, Van de Velde M, Raeder J. Active perioperative patient warming using a self-warming blanket (BARRIER EasyWarm) is superior to passive thermal insulation: a multinational, multicenter, randomized trial. J Clin Anesth. 2016 Nov;34:547-54. doi: 10.1016/j.jclinane.2016.06.030. Epub 2016 Jul 17. PMID 27687449
- [Background] Vanni SM, Braz JR, Modolo NS, Amorim RB, Rodrigues GR Jr. Preoperative combined with intraoperative skin-surface warming avoids hypothermia caused by general anesthesia and surgery. J Clin Anesth. 2003 Mar;15(2):119-25. doi: 10.1016/s0952-8180(02)00512-3. PMID 12719051
- [Background] Jo YY, Chang YJ, Kim YB, Lee S, Kwak HJ. Effect of Preoperative Forced-Air Warming on Hypothermia in Elderly Patients Undergoing Transurethral Resection of the Prostate. Urol J. 2015 Nov 14;12(5):2366-70. PMID 26571323
- [Background] Sessler DI, Schroeder M, Merrifield B, Matsukawa T, Cheng C. Optimal duration and temperature of prewarming. Anesthesiology. 1995 Mar;82(3):674-81. doi: 10.1097/00000542-199503000-00009. PMID 7879936

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convective Pre-warming | Standard of Care
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convective Pre-warming | Standard of Care | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (19) | 69.5 (2.4) | 63.7 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30 (5.7) | 33.7 (12.1) | 30.9 (8.5)
American Society of Anesthesiologists (ASA) Physical Status Classification (PS Class) [Count of Participants; unit: Participants] — ASA PS Class 2 patients were patients with mild systemic disease, while ASA PS Class 3 patients were patients with severe systemic disease.
  Participants
    ASA PS Class 2 | 4 | 3 | 7
    ASA PS Class 3 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Core Body Temperature
Description: Change in core temperature between induction of anesthesia and end of skin preparation
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Convective Pre-warming | Standard of Care
Number analyzed (Participants) | 6 | 4
Degrees Celsius | -0.95 (0.69) | -0.53 (0.85)

2. Secondary Outcome: Skin Temperature
Description: Change in skin temperature between arrival to the holding area and departure to the operating room, and arrival to the PACU
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Convective Pre-warming | Standard of Care
Number analyzed (Participants) | 6 | 4
Degrees Celsius
  Holding area to operating room departure | -0.03 (0.39) | 0.08 (0.42)
  Holding area to arrival in PACU | -0.07 (0.67) | -0.48 (0.56)

3. Secondary Outcome: Intraoperative Temperatures
Description: Core body temperature measured intraoperatively
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Convective Pre-warming | Standard of Care
Number analyzed (Participants) | 6 | 4
Degrees Celsius | 36.0 (0.79) | 35.7 (0.17)

4. Secondary Outcome: Temperature Differences Between Different Age Groups
Description: Differences in temperature changes between elderly (≥ 65 years) and younger patients (< 65 years).
Time Frame: Day 1
Population: In the Standard of care group there were only patients aged 65 years and older. This group also did not receive prewarming aside from blankets, therefore temperature was only recorded once in the preoperative unit.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Convective Pre-warming | Standard of Care
Number analyzed (Participants) | 6 | 4
Degrees Celcius
  Temperature before prewarming - Patients <65 years of age: number analyzed (Participants) | 3 | 0
  Temperature before prewarming - Patients <65 years of age | 36.5 (0.2) |
  Temperature before prewarming - Patients >65 years of age: number analyzed (Participants) | 3 | 4
  Temperature before prewarming - Patients >65 years of age | 36.6 (0.6) | 36.5 (0.4)
  Temperature after prewarming - Patients <65 years of age: number analyzed (Participants) | 3 | 0
  Temperature after prewarming - Patients <65 years of age | 36.5 (0.3) |
  Temperature after prewarming - Patients >65 years of age: number analyzed (Participants) | 3 | 0
  Temperature after prewarming - Patients >65 years of age | 36.4 (0.5) |

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Convective Pre-warming | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
Early termination due to low subject recruitment leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03876808/Prot_SAP_000.pdf